CLINICAL TRIAL: NCT06573736
Title: Stockholm3 Use Prior to MRI for Prostate Cancer Detection in a Clinical Care Pathway: a Multi-centered Validation
Acronym: S3M-MRI
Status: Not yet recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Henrik Grönberg, Professor, Karolinska Institutet
Other Study IDs: 2023-06092-01
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Stockholm3 — Stockholm3 combines protein markers tPSA, fPSA, KLK2, PSP94 and GDF15, genetic markers and clinical data to estimate risk for clinically significant prostate cancer.

SUMMARY:
Men meeting local clinical standard of care to undergo a prostate MRI for suspicion of prostate cancer will be included. Blood sample will be drawn on the day of MRI or immediately prior to MRI for measurement of the prostate cancer biomarker Stockholm3. Specifically, the Stockholm3 test will be performed in a retrospective manner and no clinical decisions will be made based on the results. The patients will not receive the results of the Stockholm3 assay. A Stockholm3 score will be reported for each patient.

The primary aim is to show superior specificity of Stockholm3 (at different thresholds) for MRI selection compared to PSA (at different thresholds) (I.e., the proportion of men with a negative Stockholm3 test or a negative PSA test among those with a normal MRI).

Additional aims:

1. To show non-inferior relative sensitivity in detection of csPC of Stockholm3 compared to PSA (The proportion of men with a positive Stockholm3 test (at different thresholds) or a positive PSA test (at different thresholds) among those diagnosed with csPC will be calculated).
2. To evaluate Stockholm3 risk thresholds to determine if it can be used to further reduce MRI, biopsy and Gleason grade group 1 cancers without reducing sensitivity of csPC detection.

ELIGIBILITY:
Inclusion Criteria:

* Men with age range (40.0 - 80.0 years)
* Already scheduled to undergo MRI for prostate cancer screening (both negative and positive MRI included).

Exclusion Criteria:

* PSA < 1.5 ng/mL
* Any known diagnosis of prostate cancer (patient on active surveillance)
* Men that have undergone digital rectal exam (DRE) immediately before blood draw (DRE within 5 days of study blood draw are excluded).
* Men who in the three (3) months prior to study participation received any invasive urologic procedure such as thermotherapy, microwave therapy, laser therapy, transurethral resection of the prostate (TURP), urethral catheterization, and lower genitourinary tract endoscopy (cystoscopy)
* No history of new treatment for BPH in three (3) months prior to study participation.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men meeting local standard of care to undergo prostate MRI for suspicion of prostate cancer
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Abnormal MRI | From enrollment up to 24 weeks
  PIRADS ≥3

SECONDARY OUTCOMES:
Clinically significant prostate cancer | From enrollment up to 24 weeks
  Grade group ≥2 prostate cancer